CLINICAL TRIAL: NCT03392584
Title: Detection and Inflammatory Characterization of Deep Infection After Surgery for Locally Advanced Rectal Cancer With Microdialysis Catheters
Status: Completed | Type: Observational
Sponsor: Oslo University Hospital (Other)
Collaborators: University of Oslo (Other)
Responsible Party: Principal Investigator, Ebbe Billmann Thorgersen, Principal Investigator, Oslo University Hospital
Other Study IDs: 2016/865
Record Dates: First submitted 2017-12-18; First posted 2018-01-08 (Actual); Last update posted 2023-04-03 (Actual); Status verified 2023-03

CONDITIONS: Locally Advanced Rectal Cancer; Abdominoperineal Resection; Infection
Keywords: Locally advanced rectal cancer; Deep infection; Microdialysis; Surgical site infection
MeSH Terms: conditions — Infections; Surgical Wound Infection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Microdialysis samples 6-10 times every day. Regularly standard blood samples. Daily samples from pelvic drain. EDTA plasma 3 times a week.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- APR: Patients with locally advanced rectal cancer treated with neoadjuvant (chemo-) radiotherapy (CRT) and operated with abdominoperineal resection (APR)
- APR with VRAM: Patients with locally advanced rectal cancer treated with neoadjuvant (chemo-) radiotherapy (CRT) and operated with abdominoperineal resection (APR) and subsequent reconstruction of the perineum with a vertical rectus abdominis myocutaneous flap (VRAM)

SUMMARY:
The intention of the study is to explore metabolic and inflammatory parameters in the pelvis after abdominoperineal resection for locally advanced rectal cancer in patients that have received radiation therapy before surgery.

DETAILED DESCRIPTION:
Locally advanced rectal cancers (LARC) threaten the normal surgical margins and therefore needs neoadjuvant (chemo-) radiotherapy to down-stage the tumor before surgery. The Norwegian Radium Hospital Oslo University Hospital is a regional center for treatment of LARC in the south-eastern part of Norway and treat approximately 80-100 patients in this category annually. About 50 of these patients receive abdominoperineal resection (APR) as the main surgical treatment. A very high rate of deep surgical site infections is reported in the APR group internationally, particularly in the patients that have received chemo-radiotherapy. The knowledge of why these patients have such a high rate of infections is scarce.

Microdialysis is a technique which enables close to real-time monitoring of the tissues and organs of interest.

The investigators want to utilize the microdialysis method to describe and monitor metabolic and inflammatory parameters, after extensive oncological surgery for LARC in patients that have undergone chemoradiotherapy before surgery. With the knowledge of how the normal biology is, the investigators hypothesize that infection can be readily detected by the biomarkers retrieved by microdialysis.

ELIGIBILITY:
Inclusion Criteria:

* Patients with primary rectal adenocarcinoma that have received radiation ≥25 Gy to the pelvis.
* operation with APR.
* have accepted and signed the consent form.

Exclusion Criteria:

* APR for other reasons

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with locally advanced rectal cancer who receive radiotherapy >25 Gy prior to surgery.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2016-10-01 (Actual); Primary Completion 2021-03-01 (Actual); Study Completion 2022-01-08 (Actual)

PRIMARY OUTCOMES:
Monitoring intermediate metabolites in the remnant muscular tissue of the pelvis floor with microdialysis catheters after neoadjuvant CRT and subsequent APR for LARC. | August 2023
  Lactate (mM), pyruvate (µM), lactate/pyruvate ratio, glycerol (µM) and glucose (mM) will be measured in microdialysis fluid from catheters inserted in the remnant muscular tissue of the pelvis floor after neoadjuvant CRT and subsequent APR for LARC to detect deep pelvic surgical site infection. The results will be compared to current standard monitoring. The measures will be done bedside on Iscus analyzer, M Dialysis AB, Stockholm, Sweden. The Iscus analyzer will calculate the lactate/pyruvate ratio.

SECONDARY OUTCOMES:
Monitoring inflammatory mediators in the remnant muscular tissue of the pelvis floor with microdialysis catheters after neoadjuvant CRT and subsequent APR for LARC. | August 2023
  Microdialysis fluid will be analysed using a multiplex cytokine assay (Bio-Plex Human Cytokine 27-Plex Panel, Bio-Rad Laboratories Inc., Hercules, CA). The following cytokines, chemokines and growth factors will be measured (all in pg/mL): Activated complement component 5 (C5a), Interleukin (IL) 1 beta (IL-1β), IL-1 receptor antagonist (IL-1Ra), IL-2, IL-4, IL-5, IL-6, IL-7, IL-8 (CXCL8), IL-9, IL-10, IL-12p70, IL-13, IL-15, IL-17, Eotaxin (CCL11), basic fibroblast growth factor (bFGF), granulocyte colony-stimulating factor (G-CSF), granulocyte-macrophage colony-stimulating factor (GM-CSF), interferon gamma (IFNG), interferon gamma inducible protein-10 (IP-10 or CXCL10), monocyte chemoattractant protein-1 (MCP-1 or CCL2), macrophage inflammatory protein-1-alpha (MIP-1α or CCL3), macrophage inflammatory protein-1-beta (MIP-1β or CCL4), platelet-derived growth factor-BB (PDGF-BB), regulated upon activation, normal T cell expressed and secreted (RANTES or CCL5), TNF-α and VEGF.
Monitoring inflammatory mediators in blood after neoadjuvant CRT and subsequent APR for LARC. | August 2023
  Blood be analysed using a multiplex cytokine assay (Bio-Plex Human Cytokine 27-Plex Panel, Bio-Rad Laboratories Inc., Hercules, CA). The following cytokines, chemokines and growth factors will be measured (all in pg/mL): Activated complement component 5 (C5a) Interleukin (IL) 1 beta (IL-1β), IL-1 receptor antagonist (IL-1Ra), IL-2, IL-4, IL-5, IL-6, IL-7, IL-8 (CXCL8), IL-9, IL-10, IL-12p70, IL-13, IL-15, IL-17, Eotaxin (CCL11), basic fibroblast growth factor (bFGF), granulocyte colony-stimulating factor (G-CSF), granulocyte-macrophage colony-stimulating factor (GM-CSF), interferon gamma (IFNG), interferon gamma inducible protein-10 (IP-10 or CXCL10), monocyte chemoattractant protein-1 (MCP-1 or CCL2), macrophage inflammatory protein-1-alpha (MIP-1α or CCL3), macrophage inflammatory protein-1-beta (MIP-1β or CCL4), platelet-derived growth factor-BB (PDGF-BB), regulated upon activation, normal T cell expressed and secreted (RANTES or CCL5), TNF-α and VEGF.
Measure inflammatory mediators in pelvic drain fluid after neoadjuvant CRT and subsequent APR for LARC. | August 2023
  Pelvic drain fluid will be analysed using a multiplex cytokine assay (Bio-Plex Human Cytokine 27-Plex Panel, Bio-Rad Laboratories Inc., Hercules, CA). The following cytokines, chemokines and growth factors will be measured (all in pg/mL): Activated complement component 5 (C5a), Interleukin (IL) 1 beta (IL-1β), IL-1 receptor antagonist (IL-1Ra), IL-2, IL-4, IL-5, IL-6, IL-7, IL-8 (CXCL8), IL-9, IL-10, IL-12p70, IL-13, IL-15, IL-17, Eotaxin (CCL11), basic fibroblast growth factor (bFGF), granulocyte colony-stimulating factor (G-CSF), granulocyte-macrophage colony-stimulating factor (GM-CSF), interferon gamma (IFNG), interferon gamma inducible protein-10 (IP-10 or CXCL10), monocyte chemoattractant protein-1 (MCP-1 or CCL2), macrophage inflammatory protein-1-alpha (MIP-1α or CCL3), macrophage inflammatory protein-1-beta (MIP-1β or CCL4), platelet-derived growth factor-BB (PDGF-BB), regulated upon activation, normal T cell expressed and secreted (RANTES or CCL5), TNF-α and VEGF.
Measure the common innate immune defect MBL deficiency in blood in the study population. | August 2023
  Measure MBL (ng/mL) in serum by an enzyme immunoassay. Compare differences in the frequency of MBL-deficiency in patients with or without deep pelvic infections.
Measure intermediate metabolites and inflammatory mediators after neoadjuvant CRT and subsequent APR for LARC with reconstruction of the perineum with VRAM. | August 2023
  Measure the above mentioned parameters and evaluate whether reconstruction with VRAM contribute to differences in these in patients after neoadjuvant CRT and subsequent APR for LARC, in comparison with patients without VRAM reconstruction.

CONTACTS AND LOCATIONS:
Overall Officials: Ebbe B Thorgersen, MD PhD, Principal Investigator — Surgeon, The Department of Gastroenterological Surgery, The Norwegian Radium Hospital, Oslo University Hospital
Locations (1):
- The Norwegian Radium Hospital Oslo University Hospital, Oslo, Norway